CLINICAL TRIAL: NCT06623734
Title: Liver CAncer PRognosis InvEstigation Study (Liver-CARE)
Brief Title: Liver Cancer Prognosis Investigation Study
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Aiping Fang, Associate Professor, Sun Yat-sen University
Other Study IDs: SYSU SPH MEC 2024-101
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Liver Neoplasms
Keywords: Primary liver cancer; Hepatocellular carcinoma; Intrahepatic cholangiocarcinoma; Prognosis; Prospective cohort study
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — liver tissues, blood, urine, and stools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This prospective cohort study is designed to explore the role of environmental, clinical, and genetic risk factors in the progression and prognosis of primary liver cancer (PLC). We will recruit 5000 patients with newly diagnosed, previously untreated PLC. The eligible patients will be asked to complete a baseline survey at the time of initial admission and be followed up every 3 to 6 months after discharge.

DETAILED DESCRIPTION:
Primary liver cancer (PLC) is highly malignant and is particularly prevalent in China. Multiple factors are involved in the development and progression of PLC. Several large-scale, prospective cohort studies have been established to identify environmental and genetic risk factors for the development of PLC in the general population. However, few cohort studies have focused on determining risk factors beyond clinical prognostic factors for the progression of PLC in patients with PLC. Therefore, we will conduct a prospective cohort study to examine the role of environmental, clinical, and genetic risk factors in the progression and prognosis of PLC. We plan to recruit 5000 patients with newly diagnosed, previously untreated PLC. A baseline survey will be conducted at the time of initial admission, with follow-up at 3 and 6 months after discharge for all patients and thereafter every 3 months for patients treated with interventional therapy and every 6 months for patients receiving surgery and other therapies. We will collect information on patients' demographics characteristics, clinical diagnosis and treatment, lifestyle, nutritional status, psychological and mental status, quality of life, anthropometric data, body composition, routine laboratory tests and examinations, and disease progression through structured questionnaires, physical examinations, and medical record reviews. Deaths will be ascertained through medical records, death certificates, and next-of-kin. Additionally, we will collect blood, urine, stool, and liver tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years,
* Diagnosed with primary liver cancer (ICD-10: C22) (Referring to the diagnostic criteria in the "Primary Liver Cancer Diagnosis and Treatment Guidelines (2024 Edition)" and the "2024 CSCO Guidelines for the Diagnosis and Treatment of Biliary Malignancies),
* Have not received any anti-tumor treatment (e.g., surgery, ablation, interventional therapy, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc),
* Signed informed consent.

Exclusion Criteria:

* Have a history of other malignant tumors,
* Have a history of other serious chronic diseases (e.g., heart failure, liver failure, kidney failure, etc.),
* Expected survival time is no more than 3 months,
* Severe physical or mental disability.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly diagnosed with primary liver cancer
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2039-12-31 (Estimated); Study Completion 2044-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | Up to 20 years
  The primary endpoint of this study is all-cause mortality and liver caner-specific mortality. The exact death time and the cause of death of each participant will be checked in the government medical records system.

SECONDARY OUTCOMES:
Recurrence (intrahepatic and extrahepatic) | From date of diagnosis until the date of cancer recurrence or date of death from any cause, whichever came first, assessed up to 20 years
  Time of recurrence will be obtained by telephone interview or medical treatment records
Newly Emerging Diseases | From date of diagnosis until the date of newly emerging diseases or date of death from any cause, whichever came first, assessed up to 20 years
  Time of newly emerging diseases will be obtained by telephone interview or medical treatment records
Response Evaluation | through study period, every 3-6 months
  For patients undergoing surgical treatment, assess whether there is recurrence. For patients receiving ablation therapy, evaluate whether the tumor is completely ablated. For patients undergoing interventional therapy and radiotherapy, use the modified Response Evaluation Criteria in Solid Tumors (mRECIST) for hepatocellular carcinoma to evaluate efficacy. Use the RECIST 1.1 criteria for efficacy evaluation for patients undergoing systemic anticancer treatment. For patients receiving anti-angiogenic molecular targeted therapy, use the mRECIST criteria in combination. For patients receiving immuno-checkpoint inhibitor therapy, use the iRECIST criteria. Short-term efficacy evaluation indicators include the objective response rate (ORR), progression-free survival (PFS), disease-free survival (DFS), etc.
Nutritional status | through study period, every 3-6 months
  To assess the nutritional risk, the patient will be screened by Nutrition Risk Screening 2002 (NRS-2002), patient-generated subjective global assessment (PG-SGA), the global leadership initiative on malnutrition (GLIM).
Quality of life | through study period, every 3-6 months
  The assessment is based on the European Organization for Research and Treatment of Cancer (EORTC) quality of life core questionnaire QLQ-C30 for all cancer patients, the specific quality of life subscale QLQ-HCC18 for patients with liver cancer or QLQ-BIL21 for patients with intrahepatic cholangiocarcinoma.
Psychological and mental status | through study period, every 3-6 months
  Anxiety and depression are evaluated using the Generalized Anxiety Disorder 7-item scale (GAD-7) and Patient Health Questionnaire 9-item Depression Scale (PHQ-9), recommended by the American Society of Clinical Oncology (ASCO) Adult Cancer Survivor Anxiety and Depression Management Guidelines.
Cachexia assessment | through study period, every 3-6 months
  Use the Anorexia Cachexia Subscale-12 (A/CS-12) to assess anorexia, and utilize the CASC-IN tool to evaluate whether the patient has cachexia. If cachexia is present, the cachexia scoring system (CASCO) should be used for further assessment of the cachexia stage.
Sarcopenia | through study period, every 3-6 months
  Utilize the Simple Five-Item Scale (SARC-F) questionnaire to screen if the study subjects have sarcopenia.
Frailty | through study period, every 3-6 months
  Assess frailty using the Liver Frailty Index (LFI). This index considers the following assessment items: (1) Dominant hand grip strength; (2) Time to do 5 chair stands; and (3) Seconds holding 3 position balance.

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Fang, MBBS, PhD, Principal Investigator — Sun Yat-sen University; Yanjun Zhang, MBBS, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No